CLINICAL TRIAL: NCT00981903
Title: Tinzaparin for Primary Treatment and Extended Secondary Prophylaxis of Venous Thromboembolism in Patients With Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Tinzaparin will no longer be available in the United States
Sponsor: University of Southern California (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0S-04-5
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Venous Thromboembolism; Cancer
Keywords: VTE in cancer patients
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VTE Treatment Group (Experimental)
  Interventions: Drug: Tinzaparin sodium
- Control (No Intervention)

INTERVENTIONS:
Drug: Tinzaparin sodium — Subcutaneous injection 175 U/Kg/day
  Arms: VTE Treatment Group

SUMMARY:
In this study the investigators will determine the safety and effectiveness of Tinzaparin in preventing blood clots for up to 12 months of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to use long-term administration of a low molecular weight heparin (tinzaparin) for primary treatment and secondary prophylaxis of venous thromboembolism in patients with cancer. We will determine the efficacy (recurrent VTE) and safety (major hemorrhage) of this approach. Secondarily, we will analyze the outcome of patients in terms of survival and response to therapy versus matched controls. We will also determine baseline levels of markers of hemostasis, fibrinolysis, and angiogenesis and will follow changes with treatment as well as correlate levels of these plasma markers with outcomes, including recurrent venous thromboembolism, major hemorrhage,and survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active cancer
* Patients have documented or recurrent malignancy and must meet at least one of the following criteria:

  * Diagnosis or documented presence of cancer within 6 months, excluding squamous cell or basal cell carcinoma of the skin OR
  * Receive any therapy for cancer within the previous 6 months OR
  * Currently receiving any treatment (surgery, radiation, chemotherapy, hormonal therapy, biotherapy, palliative therapy, and/or combined modality therapy) for cancer
* Documented first venous thromboembolic event
* Patients must meet at least one of the following criteria:

  * Deep vein thrombosis of the lower extremity confirmed with duplex ultrasonography, magnetic resonance imaging, or venogram OR
  * Pulmonary embolism confirmed with high probability V/Q scan, CT angiogram, or pulmonary angiogram
* ECOG performance status of 0, 1, or 2
* Signed written informed consent
* Age 18 years or greater

Exclusion Criteria:

* Body weight less than 40 kg
* Recurrent spontaneous fractures unrelated to the underlying active malignancy
* Administration of therapeutic doses of unfractionated or low molecular weight heparin for more than 48 hours prior to registration Amendment 3 (05/26/2009) 11
* Need for long-term oral anticoagulant therapy (e.g., mechanical heart valves, atrial fibrillation)
* Poor performance status with an ECOG score of 3 or 4
* Serious hemorrhage requiring hospitalization, transfusion, or surgical intervention within 2 weeks of presentation
* Known acute (symptomatic or active bleeding) gastroduodenal ulcer
* Epidural/spinal puncture within the last 24 hours
* Neurosurgery within 1 week of registration or any previous history of intracranial hemorrhage
* Septic endocarditis
* Overt pericardial effusion
* Current platelet count of less than 50 x 109/L
* Undergoing high dose chemotherapy for peripheral blood stem cell or bone marrow transplantation, induction chemotherapy for acute leukemia, or has other conditions associated with persistent thrombocytopenia of less than 100 109/L for a duration of at least four consecutive weeks
* Familial bleeding diathesis
* Uncontrolled hypertension despite antihypertensive therapy
* Dependent upon renal dialysis or significant renal failure with a serum creatinine of greater than three times the upper limit of normal
* Allergy to heparin (unfractionated or low molecular weight)
* Allergy to contrast medium
* Pregnant or of childbearing potential and not using adequate contraception
* Geographically inaccessible for follow-up
* Failure or inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-07; Primary Completion 2012-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Development of recurrent venous thromboembolism and major hemorrhage. | up to 6 months on treatment

SECONDARY OUTCOMES:
Secondary outcome measures will evaluate other thrombotic events, clinical cancer outcome, and plasma markers of hemostasis, fibrinolysis, and angiogenesis | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Cornell Weill Scholl of Medicine, New York, New York